CLINICAL TRIAL: NCT03229980
Title: Pediatric Myocardial Protection; Large Volume Potassium Cardioplegia Advantageous Over Small Volume Potassium Cardioplegia: Where do we Stand?
Brief Title: Pediatric Myocardial Protection With Potassium Cardioplegia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sayed Kaoud Abd-Elshafy, Associate Profossor of Anesthesiology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00008715918
Record Dates: First submitted 2017-07-23; First posted 2017-07-26 (Actual); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Cardioplegia
Keywords: myocardial protection; potassium cardioplegia; tropinin; Custodiol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group L (Active Comparator): Hearts will be arrested with cold blood cardioplegia, first dose (arrest dose) will be 30 ml/kg and the frequent doses every 20 min will be 15 ml/kg The content of cardioplegic solution will be (K+, 10mmol/L) lidocaine 50 mg/L, magnesium sulphate 1 gm/L,dextrose 25% 25 mL/L and sodium bicarbonate 8.4% 25 mL/L during cardiac surgery. Cardioplegic infusion duration will be infused over 300s.
  Interventions: Drug: Cold blood cardioplegia (large volume)
- Group S (Active Comparator): Hearts will be arrested with cold blood cardioplegia first dose (arrest dose) will be 10 ml/kg and the frequent doses every 20 min will be 5 ml/kg The content of cardioplegic solution will be (K+, 30mmol/L) lidocaine 150 mg/L, magnesium sulphate 3 gm/L, dextrose 25% 25 mL/L and sodium bicarbonate 8.4% 25 mL/L during cardiac surgery.
  Interventions: Drug: Cold blood cardioplegia (small volume)

INTERVENTIONS:
Drug: Cold blood cardioplegia (large volume) — Hearts will be arrested with cold blood cardioplegia, first dose (arrest dose) will be 30 ml/kg and the frequent doses every 20 min will be 15 ml/kg
  Arms: Group L
Drug: Cold blood cardioplegia (small volume) — Hearts will be arrested with cold blood cardioplegia first dose (arrest dose) will be 10 ml/kg and the frequent doses every 20 min will be 5 ml/kg
  Arms: Group S

SUMMARY:
The advances in cardiac surgery and anesthesia for pediatric patients planned for repair of congenital heart disease encourage us to discuss problems that occur during this surgery especially during Cardiopulmonary Bypass (CPB). Cardiopulmonary Bypass induces a damaging systemic inflammatory response, in addition to a myocardial ischemia-reperfusion injury (IRI) as a result of cessation and re-initiation of coronary artery circulation

DETAILED DESCRIPTION:
After approval of the local ethics committee of Assiut University and obtaining written informed consent from parents or guardians of all patients, 60 patients with congenital heart disease will be included. Patients will be randomly allocated into three groups

ELIGIBILITY:
Inclusion Criteria

* Scheduled cardiac surgery requiring cardioplegic arrest with expected cross clamp time>45 minutes.
* Hemodynamic stability.

Exclusion Criteria:

* Previous cardiac surgery.
* Urgent or emergent cases.
* Any known allergies to components of either cardioplegia solutions.

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 87 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-04-03 (Actual); Study Completion 2018-04-28 (Actual)

PRIMARY OUTCOMES:
Cardiac rhythm on return | within the first 24 hours
  Sinus rhythm or Ventricular Fibrillation:
  DC will be used or not and if used how much joules and how many times.

SECONDARY OUTCOMES:
The inotropic score | within one month
  1 point is assigned for each mcg/kg/min of dopamine and dobutamine, and 10 points is assigned for each 0.1 mcg/kg/min of epinephrine, norepinephrine, and phenylephrine. (i.e. 1 point is assigned for each 10 ng/kg/min of epinephrine, norepinephrine, and phenylephrine.
Cardiac dysrhythmias | within the first week
  Cardiac dysrhythmias during intensive care unit stay
blood pressure | within the first 24 hours
  blood pressure
transthoracic echocardiography (TTE) changes | within the first week
  Changes in ejection fraction by TTE
Troponin I levels | within the first 24 hours
  We will obtain blood samples for troponin I levels (as a marker of myocardial ischemia) pre-CBP, 6, 12 and 24 hours after the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sayed k Abd-Elshafy, MD, Principal Investigator — Associate profossor of anesthesiology
Locations (1):
- Faculty of Medicine, Asyut, Egypt